CLINICAL TRIAL: NCT03128034
Title: A Study Evaluating Escalating Doses of 211^At-Labeled Anti-CD45 MAb BC8-B10 (211^At-BC8-B10) Followed by Allogeneic Hematopoietic Cell Transplantation for High-Risk Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL), or Myelodysplastic Syndrome (MDS)
Brief Title: 211^At-BC8-B10 Before Donor Stem Cell Transplant in Treating Patients With High-Risk Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Myelodysplastic Syndrome, or Mixed-Phenotype Acute Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9595; NCI-2017-00452 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9595 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA078902 (NIH); RG9217014 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome With Excess Blasts; Recurrent Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia; Recurrent Acute Lymphoblastic Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Refractory Acute Myeloid Leukemia; Refractory Mixed Phenotype Acute Leukemia; Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts; Leukemia, Biphenotypic, Acute | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (211^At-BC8-B10, PBSC) (Experimental): Patients receive 211^At-BC8-B10 IV over 6-8 hours on day -7 and may receive 131^I-BC8-B10 IV on day -7 and fludarabine phosphate IV over 30 minutes on days -4, -3 and -2. Patients undergo TBI and PBSC transplant on day 0. Patients also receive cyclosporine PO or IV every 12 hours on days -3 to 56 and then tapered to day 180, or continuing to day 96 and then tapered to day 150. Patients receive mycophenolate mofetil PO or IV (first dose to occur 4-6 hours after PBSC infusion) every 12 hours on days 0-27 (for patients with related donors) or every 8 hours on day 0 and then reduced to every 12 hours on days 30-150 then tapered to day 180 (for patients with unrelated donors). Patients may undergo SPECT, bone marrow aspirate sample and blood sample collection on study.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Pretargeted Radioimmunotherapy; Radiation: Total-Body Irradiation; Procedure: Biospecimen Collection; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Drug: Cyclosporine — Given PO or IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Radiation: Pretargeted Radioimmunotherapy — Given 211^At-BC8-B10 IV
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation; TBI; Whole Body Irradiation; SCT_TBI
Radiation: Pretargeted Radioimmunotherapy — Given 131^I-BC8-B10 IV
Procedure: Biospecimen Collection — Undergo blood and bone marrow aspirate sample collection
  Other Names: Biological Sample Collection
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT
  Other Names: SPECT; SPECT SCAN; Medical Imaging

SUMMARY:
This phase I/II trial studies the side effects and best dose of 211^astatine(At)-BC8-B10 before donor stem cell transplant in treating patients with high-risk acute myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome, or mixed-phenotype acute leukemia. Radioactive substances, such as astatine-211, linked to monoclonal antibodies, such as BC8, can bind to cancer cells and give off radiation which may help kill cancer cells and have less of an effect on healthy cells before donor stem cell transplant.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of 211^At-BC8-B10.

Patients receive 211^At-BC8-B10 intravenously (IV) over 6-8 hours on day -7 and may receive 131^I-BC8-B10 IV on day -7 and fludarabine phosphate IV over 30 minutes on days -4, -3 and -2. Patients undergo TBI and peripheral blood stem cell (PBSC) transplant on day 0. Patients also receive cyclosporine orally (PO) or IV every 12 hours on days -3 to 56 and then tapered to day 180 (for patients with related donors), or continuing to day 96 and then tapered to day 150 (for patients with unrelated donors). Patients receive mycophenolate mofetil PO or IV (first dose to occur 4-6 hours after PBSC infusion) every 12 hours on days 0-27 (for patients with related donors) or every 8 hours on day 0 and then reduced to every 12 hours on days 30-150 then tapered to day 180 (for patients with unrelated donors). Patients may undergo single photon emission computed tomography (SPECT), bone marrow aspirate sample and blood sample collection on study.

After completion of study treatment, patients are followed up at 100 days and then at 6, 9, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have AML, ALL, high-risk MDS, or MPAL (also known as biphenotypic) meeting one of the following descriptions:

  * AML, ALL, or MPAL in first remission with evidence of measurable residual disease (MRD) by flow cytometry
  * AML, ALL, or MPAL beyond first remission (i.e., having relapsed at least one time after achieving remission in response to a treatment regimen)
  * AML, ALL, or MPAL representing primary refractory disease (i.e., having failed to achieve remission at any time following one or more prior treatment regimens)
  * AML evolved from myelodysplastic or myeloproliferative syndromes
  * MDS expressed as refractory anemia with excess blasts (RAEB)
  * Chronic myelomonocytic leukemia (CMML) by French-American-British (FAB) criteria
* Patients not in remission must have CD45-expressing leukemic blasts. Patients in remission do not require phenotyping and may have leukemia previously documented to be CD45 negative (because in remission patients, virtually all antibody binding is to non-malignant cells which make up >= 95% of nucleated cells in the marrow)
* Patients must be >= 18 and =< 75 years of age
* Patients should have a circulating blast count of less than 10,000/mm^3 (control with hydroxyurea or similar agent is allowed)
* Patients must have an estimated creatinine clearance greater than 50/ml per minute by the following formula (Cockcroft-Gault); serum creatinine value must be within 28 days prior to registration
* Patients must have normal hepatic function (bilirubin within normal limits, aspartate aminotransferase [AST] and alanine aminotransferase [ALT] < 2 times the upper limit of normal) within 2 months prior to the astatine-211 infusion date (with the exception of patients that are known to have Gilbert's disease, for whom total bilirubin is allowed up to 3 x upper limit of normal [ULN])
* Eastern Cooperative Oncology Group (ECOG) < 2 or Karnofsky >= 70
* Patients must be free of uncontrolled infection
* Patients with prior non-myeloablative or reduced-intensity conditioning allogeneic-hematopoietic cell transplant (HCT) must have no evidence of ongoing GVHD and be off GVHD treatment immunosuppression for at least 6 weeks at time of enrollment
* Patients must have normal elastography
* If ferritin is elevated, patient must have less than 7 mg/g liver iron concentration on liver T2* MRI
* Patients should have an official gastrointestinal (GI) consult prior to the transplant for full evaluation
* Patients must have an HLA-matched related donor or an HLA-matched unrelated donor who meets standard Fred Hutch and/or National Marrow Donor Program (NMDP) or other donor center criteria for peripheral blood stem cell (PBSC) or bone marrow donation, as follows:

  * Related donor: related to the patient and genotypically or phenotypically identical for HLA-A, B, C, DRB1 and DQB1; phenotypic identity must be confirmed by high-resolution typing
  * Unrelated donor:

    * Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; OR
    * Mismatched for a single allele without antigen mismatching at HLA-A, B, or C as defined by high resolution typing but otherwise matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
    * Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results; a positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
  * Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed

Exclusion Criteria:

* Patients may not have symptomatic coronary artery disease and may not be on cardiac medications for anti-arrhythmic or inotropic effects
* Left ventricular ejection fraction < 35%
* Corrected diffusing capacity of the lungs for carbon monoxide (DLCO) < 35% or receiving supplemental continuous oxygen; when pulmonary function test (PFT)s cannot be obtained, the 6-minute walk test (6MWT, also known as exercise oximetry) will be used: Any patient with oxygen saturation on room air of < 89% during a 6MWT will be excluded
* Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease
* Patients who are known to be seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures
* Active central nervous system (CNS) leukemia at time of treatment
* Patients with prior myeloablative allogeneic-HCT
* Women of childbearing potential who are pregnant (beta-human chorionic gonadotropin positive [beta-HCG+] or breast feeding
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant
* Inability to understand or give an informed consent
* Allergy to murine-based monoclonal antibodies
* Known contraindications to radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grades III/IV Bearman regimen-related toxicity | Up to 100 days following hematopoietic cell transplantation
  The maximum tolerated dose will be defined as the dose of 211^At-BC8-B10 used in combination with the reduced-intensity hematopoietic cell transplantation conditioning regimen that is associated with a grade III/IV regimen-related toxicity or true dose limiting toxicity rate of 25%.the data, thereby generating a dose-response curve based on the observed toxicity rate at the various dose levels visited. Based on this fitted model, the maximum tolerated dose is estimated to be the dose that is associated with a toxicity rate of 25%.

SECONDARY OUTCOMES:
Engraftment | Up to day 100
  Sufficient evidence will be taken to be a lower limit of the appropriate 80% one-sided confidence interval associated with the estimated proportion of rejections in excess of 0.20.
Chimerism | Up to day 84
Non-relapse mortality | Up to 2 years
Acute graft versus host disease | Up to day 180
Achievement of remission | Up to 2 years
Duration of remission | Up to 2 years
Overall survival | Up to 100 days
Disease-free survival | Up to 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Brenda M. Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Li Y, Hamlin DK, Chyan MK, Wong R, Dorman EF, Emery RC, Woodle DR, Manger RL, Nartea M, Kenoyer AL, Orozco JJ, Green DJ, Press OW, Storb R, Sandmaier BM, Wilbur DS. cGMP production of astatine-211-labeled anti-CD45 antibodies for use in allogeneic hematopoietic cell transplantation for treatment of advanced hematopoietic malignancies. PLoS One. 2018 Oct 18;13(10):e0205135. doi: 10.1371/journal.pone.0205135. eCollection 2018. PMID 30335787